CLINICAL TRIAL: NCT01901003
Title: SEDATIVE PREMEDICATION: EFFICACY ON PATIENT EXPERIENCE
Acronym: PremedX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-005171-16; 2011-32 (Other: AP HM)
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Perioperative Anxiety
MeSH Terms: interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo group (Placebo Comparator): placebo
  Interventions: Drug: Placebo (microcrystalline celluloses)
- no premedication group (Active Comparator): no premedication
  Interventions: Other: no premedication
- Lorazepam group (Experimental): lorazepam
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam
  Arms: Lorazepam group
Other: no premedication
  Arms: no premedication group
Drug: Placebo (microcrystalline celluloses)
  Arms: placebo group

SUMMARY:
Seven French university hospitals will participate in this multicentric prospective, blinded and randomized study. The investigators designed 3 study groups: Lorazepam 2.5mg, Placebo (microcrystalline celluloses) and no premedication at all. The third group (no premedication) is necessary in order to evaluate a placebo response, which may be significant on anxiety level and patients perceptions of care. It was calculated that 969 patients had to be included in order to obtain a 5 point difference between groups on the EVAN score with 80 % statistical power, leading to the inclusion of 1200 patients with an estimated maximum dropout rate of 15 %. All adults below 70 years and scheduled for elective surgery under general anesthesia can be included after information by an anesthesiologist in charge of the study and written informed consent. Non inclusion criterions are: a weight below 45 Kg, a counter indication to benzodiazepine, surgeries that could impair cognitive functions (cardiac or neurologic surgery), usual use of neuroleptics or lithium, drug addiction or former cognitive disease. The technique of anesthesia will be decided by the attending anesthesiologist, who will be unaware of the premedication technique, independently of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18 to 70 years or more;
* About a weight greater than 45 kg;
* Subject to benefit from a scheduled surgery under general anesthesia;
* Topic respecting the ambivalence clause defined below:

  1. Having no cons-indication to the use of benzodiazepines;
  2. Having no known allergy to benzodiazepines;
  3. May be a candidate for the prescription of premedication;
* Topic able to complete a self-administered questionnaire;
* Subject has signed a written informed consent and agreeing to abide by the instructions of the Protocol

Exclusion Criteria:

* - Topic of over 70 years;
* Topic 45 kg or less;
* Topic demanding to receive anxiolytic premedication;
* Subject severe respiratory insufficiency;
* Topic minor, pregnant or breastfeeding, about not being affiliated to the social security system;
* Topic for which surgery is performed under local anesthesia;
* Subject unable to perform only a self-administered questionnaire (inability to read French, severe cognitive impairment);
* Subject to which the scheduled surgery may cause postoperative cognitive dysfunction (intracranial surgery, extracorporeal circulation);
* Topic scheduled for obstetrical surgery or outpatient;
* Subject treated with antipsychotic (neuroleptic or lithium);
* Subject with cognitive impairment already documented (Alzheimer, dementia, neurological sequelae);
* Subject active consumer of narcotics;
* Subject has not signed informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the EVAN score | 2 years
  to evaluate patient satisfaction of the perioperative period

SECONDARY OUTCOMES:
the perioperative level of anxiety | 2 years
  APAIS score (Moerman 1996) before surgery

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Maurice-Szamburski A, Auquier P, Viarre-Oreal V, Cuvillon P, Carles M, Ripart J, Honore S, Triglia T, Loundou A, Leone M, Bruder N; PremedX Study Investigators. Effect of sedative premedication on patient experience after general anesthesia: a randomized clinical trial. JAMA. 2015 Mar 3;313(9):916-25. doi: 10.1001/jama.2015.1108. PMID 25734733